CLINICAL TRIAL: NCT00332748
Title: Effect of Esomeprazole on the Pharmacokinetics of BMS-275183 in Patients With Advanced Malignancies
Brief Title: A Phase I Study of BMS-275183 (Oral Taxane) Given on a Daily Schedule in Combination With Esomeprazole (Nexium) in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA165-030
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — taxane

INTERVENTIONS:
Drug: Oral Taxane

SUMMARY:
The purpose of this study is to determine what effects Esomeprazole (Nexium) has on increasing or decreasing the amount of oral taxane in the blood, and to determine the safety of oral taxane and effect of oral taxane on the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancers excluding cancers within the blood
* Adequate kidney and liver function
* > = 4 weeks from last course of chemotherapy

Exclusion Criteria:

* Inability to swallow capsules
* Other active medical disorder
* Abnormal heart function or use of drugs that affect the heart

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2006-12; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of taking Nexium in combination with oral taxane and the effect this combination has on oral taxane's exposure levels in the body.

SECONDARY OUTCOMES:
To assess the safety of a single dose of oral taxane followed by a therapeutic regimen of oral taxane administered twice weekly

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Local Institution, Newark, Delaware
  - Local Institution, Louisville, Kentucky
  - Local Institution, Las Vegas, Nevada
- Local Institution, Amsterdam, Netherlands